CLINICAL TRIAL: NCT02409316
Title: [18F]Fluoroestradiol (FES) PET/CT Imaging to Evaluate in Vivo ER in Endocrine Refractory Metastatic Breast Cancer
Brief Title: [18F]FES PET/CT in Endocrine Refractory Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 821717; NCT02559544 (obsolete NCT alias)
Record Dates: First submitted 2015-03-31; First posted 2015-04-06 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Estrogen Receptor Positive Breast Cancer; Breast Neoplasm; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 16-fluoroestradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FES PET/CT (Experimental): All subjects will receive an [18F]FES PET/CT scan.
  Interventions: Drug: [18F]FES

INTERVENTIONS:
Drug: [18F]FES — [18F]FES PET/CT scan
  Other Names: Fluoroestradiol

SUMMARY:
In this study, positron emission tomography (PET/CT) imaging will be used to evaluate estrogen receptor (ER) activity in sites of metastatic disease using the investigational radiotracer [18F]fluoroestradiol (FES).

DETAILED DESCRIPTION:
This study will evaluate [18F]FES PET/CT uptake as a predictor of progression free survival in endocrine refractory recurrent or metastatic breast cancer patients starting a new therapy regimen including endocrine targeted therapy. Imaging will occur prior to starting new therapy. Some patients may also undergo a second FES PET/CT scan at the time of suspected progression of disease to compare for changes in FES uptake measures. This is an observational study in that [18F]FES PET/CT will not be used to direct therapy decisions.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Recurrent or metastatic cancer that is of known or suspected breast origin - may be biopsy proven or identified on standard imaging (e.g. CT, bone scan, MRI, FDG PET/CT)
3. History of ER+ pathology (ER+ may be confirmed from surgery or biopsy of primary breast cancer or lymph nodes, and/or surgery or biopsy of a metastatic site, metastatic biopsy is not required)
4. At least one site of disease outside of the liver that is seen on standard imaging (e.g. CT, bone scan, MRI, FDG PET/CT); patients with measurable or nonmeasurable disease are allowed.
5. History of progression or recurrence of disease while on an endocrine targeted therapy containing regimen as assessed by medical record review of breast cancer history at screening
6. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures

Exclusion Criteria:

1. Females who are pregnant at the time of screening will not be eligible for this study, urine pregnancy test will be performed at screening in women of child-bearing potential.
2. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
3. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
4. History of HER2/neu positive cancer (IHC 3+ and/or FISH positive) as assessed by medical record review at screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-05; Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluate [18F]FES PET/CT Uptake | 4 years
  Evaluate [18F]FES PET/CT uptake as a predictor of progression free survival in endocrine refractory recurrent or metastatic breast cancer patients starting a new therapy regimen including endocrine targeted therapy

SECONDARY OUTCOMES:
Correlate [18F]FES Uptake Measures with Standard Immunohistochemistry | 4 years
  Correlate [18F]FES uptake measures with standard immunohistochemistry (IHC) (e.g. ER, PR, HER2-neu) and experimental pathology markers available from primary and/or metastatic tissue
Evaluate the utility of combined [18F]FES PET/CT and FDG PET/CT | 4 years
  Evaluate the utility of combined [18F]FES PET/CT and FDG PET/CT in identifying heterogeneity of estrogen receptor expression and functionality in metastatic breast cancer
Evaluate Overall Survival in Patients | 4 years
  Evaluate overall survival in patients receiving regimens containing endocrine targeted therapy
Compare FES Uptake Measures at Baseline and Progression | 4 years
  Compare FES uptake measures at baseline and progression in patients receiving additional endocrine targeted therapy
Correlate FES uptake measures with number of ER+ Circulating Tumor Cells | 4 years
  Correlate FES uptake measures with number of ER+ Circulating Tumor Cells (CTCs) and ratio of ER+ to ER- CTCs

CONTACTS AND LOCATIONS:
Overall Officials: David Mankoff, MD. PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Hospital, Philadelphia, Pennsylvania, United States